CLINICAL TRIAL: NCT05945654
Title: Subjective Functional Outcome After Oesophagectomy With and Without Anastomotic Leak
Brief Title: Functional Outcome After Anastomotic Leak After Oesophagectomies
Acronym: FOAL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Stefan Gutknecht (Other)
Responsible Party: Sponsor-Investigator, Stefan Gutknecht, Principal Investigator, Stadtspital Zürich
Organization: Stadtspital Zürich (Other)
Other Study IDs: BASEC 2022-01799
Record Dates: First submitted 2023-06-06; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Anastomotic Leak Esophagus; Swallowing Disorder
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anastomotic leak: Patients who had an Ivor Lewis Oesophagectomy and suffered an anastomotic leak (AL) postoperatively. AL, as defined according to ECCG (Esophagectomy Complication Consensus Group) criteria 1-3.
  Interventions: Procedure: Anastomotic Leak after Ivor Lewis Oesophagectomy
- No anastomotic leak: Patients who had an Ivor Lewis Oesophagectomy and had no AL postoperatively, ECCG 0.

INTERVENTIONS:
Procedure: Anastomotic Leak after Ivor Lewis Oesophagectomy — Surgical resection of the esophagus with oesophagogastrostomy. Groups depend on postoperative complication
  Groups: Anastomotic leak

SUMMARY:
The main surgical treatment for oesophageal cancer is a curative resection, mostly performed according to Ivor Lewis. However, despite careful work and refined surgical techniques, anastomotic leakage (AL) occurs in more than 1/10 of the patients. This severe complication normally requires immediate intervention, while over the last 10 years, endoscopic vacuum therapy (EVT) has become the crucial therapy for broken-down anastomosis. The hypothesis is that despite suffering a severe complication, the subjective swallow function is not impaired in patients treated by EVT after an anastomotic leak, compared to patients without AL.

DETAILED DESCRIPTION:
The investigators will select patients after oesophagectomy and perform a structured interview regarding their quality of life and subjective swallow function. Results will be compared according to defined subgroups, especially patients with and without anastomotic leak.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received an Ivor Lewis Oesophagectomy with reconstruction due to any reason
* Patients older than 18 years

Exclusion Criteria:

* Patients with achalasia
* inability to understand study procedure or to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients, according to the above mentioned criteria who were operated at Stadtspital Triemli between 01.06.2018 and 31.5.2022
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Swallow function by questionnaires: Sydney Swallow Questionnaire (SSQ) | earliest 6 months postoperatively
  This questionnaire consists of 17 questions and is mainly based on a visual analog scale (VAS) to assess functional swallowing. The sum of all questions ranges from 0-1700. The calculated upper limit of the reference interval is 234 in a non-dysphagic population. A higher score represents a more severe dysphagia.
Swallow function by questionnaires: Eckardt Score (ES) | earliest 6 months postoperatively
  The ES is a questionnaire with four items (weight loss, chest pain, regurgitation, and dysphagia) initially used to evaluate achalasia. The maximum score is 12; the higher the score, the more trouble patients have with swallowing.
Swallow function by questionnaires: Brief Esophageal Dysphagia Questionnaire (BEDQ) | earliest 6 months postoperatively
  The BEDQ has 10 questions to score dysphagia specifically. The questions are answered using a Likert scale (low to high), which sums up to a score ranging from 0 (asymptomatic) to 40.

SECONDARY OUTCOMES:
Quality of life by questionnaires EORTC-C30 (European Organisation for Research and Treatment of Cancer-Cancer 30) | earliest 6 months postoperatively
  The European Organisation for Research and Treatment of Cancer (EORTC) has a quality-of-life questionnaire for cancer patients. Depending on the tumor localization, a different combination of modules is used. This study combines the general 'C30' module with 30 items and the supplemental oesophagogastric 'OG25' module with 25 items.
  The transformed score of the C30 module ranges from 0 to 100. A high score represents a high level of symptomatology.
Quality of life by questionnaires EORTC-OG25 (Oesophagogastric-25) | earliest 6 months postoperatively
  As stated above, in addition to the EORTC-C30 module, the EORTC OG25 module is used. These items can be analyzed for several symptoms and are standardized by a formula to a value ranging from 0 to 100. Again a higher score represents more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Gutknecht, MD, Principal Investigator — Stadtspital Zurich
Locations (1):
- Stadtspital Zurich, Triemli, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No